CLINICAL TRIAL: NCT06052618
Title: Phase II Study of Pacritinib in Kaposi Sarcoma Herpesvirus (KSHV)-Associated Multicentric Castleman Disease and KSHV-Associated Inflammatory Cytokine Syndrome (KICS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001537; 001537-C
Record Dates: First submitted 2023-09-22; First posted 2023-09-25 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09-03

CONDITIONS: KSHV Inflammatory Cytokine Syndrome (KICS); Kaposi Sarcoma Herpesvirus -Associated Multicentric Castleman Disease
Keywords: JAK2; Interleukin-1; interleukin 6 receptor; Lymphoproliferative Disorder; HIV
MeSH Terms: conditions — Lymphoproliferative Disorders | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Treatment with pacritinib
  Interventions: Drug: Pacritinib

INTERVENTIONS:
Drug: Pacritinib — Pacritinib is administered orally as 200 mg twice daily for a total of 6, 28-day cycles

SUMMARY:
Background:

Kaposi sarcoma herpesvirus (KSHV)-associated inflammatory cytokine syndrome (KICS) and KSHV-multicentric Castleman disease (MCD) occur in people living with HIV. These diseases cause severe inflammation that can be fatal if not treated.

Objective:

To test a drug (pacritinib) in people with KSHV-associated KICS or MCD.

Eligibility:

People aged 18 years and older with KSHV-associated KICS or MCD. They must have at least one symptom.

Design:

Participants will be screened. They will have a physical exam with blood tests and tests of their heart function. They will have imaging scans. Their ability to perform everyday tasks will be reviewed. In some participants who have Kaposi sarcoma (KS) with KICS or MCD, these individuals may need a bronchoscopy and/or endoscopy of the upper or lower intestine: A flexible tube with a camera and a light source will be inserted through the mouth or anus to see these structures and assess any KS.

Pacritinib is a capsule taken by mouth. Participants will take the drug twice a day, every day, for up to 24 weeks. They will write down each dose in a diary.

Participants will visit the clinic 3 times in the first 4 weeks. Their visits will taper to once every 4 weeks. Imaging scans, blood tests, and other tests will be repeated during these visits. Participants will give samples of saliva. They may opt to allow tissues samples to be taken from their skin and lymph nodes.

Participants will have follow-up visits 7 days and 30 days after their last dose of pacritinib. After that, they will visit the clinic every 3 months for up to 1 year. The physical exam and blood, heart, and imaging tests will be repeated at these visits.

DETAILED DESCRIPTION:
Background:

* Pacritinib, is a JAK2/tyrosine kinase 3 inhibitor with negligible activity against JAK1 that also suppresses the interleukin-1 (IL-1) directed inflammatory pathway via inhibition of interleukin 1 receptor associated kinase.
* Phase III studies of patients with myelofibrosis treated with pacritinib have demonstrated safety and efficacy as compared with best available treatment.
* Pacritinib at 200mg twice daily emerged as the recommended dose in the treatment of myelofibrosis.
* Through its activity on JAK2 and IRAK1, pacritinib blocks signaling through the interleukin 6 receptor (IL-6R); this should also include signaling through gp130 mediated by KSHV vIL-6.
* In preliminary unpublished results, the Yarchoan lab has found that pacritinib is highly active against primary effusion lymphoma (PEL) cells in vitro. PEL is caused by Kaposi sarcoma associated herpesvirus (KSHV), and most PEL affected patients are co-infected with Epstein- Barr virus (EBV). Like the plasmablasts of KSHV- multicentric Castleman disease (MCD), PEL cells are KSHV-infected B cells and thus can be a model for KSHVMCD.
* Given the overlapping cytokine profile between KSHV-MCD and KSHV-associated inflammatory cytokine syndrome (KICS) and elevated levels of IL6, we expect that pacritinib will have therapeutic effect in this disorder that is associated with excess inflammation.

Objective:

-To evaluate the clinical benefit of pacritinib in participants with symptomatic KSHV-MCD or KICS using a modified KSHV-MCD/KICS Clinical Benefit Response Criteria

Eligibility:

* Pathologically confirmed MCD or evidence of KICS
* Age >= 18
* At least one clinical symptom and at least one laboratory attributable to KSHV-MCD or KICS
* ECOG performance status <= 3
* No life- or organ-threatening manifestations of MCD or KICS
* No concurrent diagnosis of PEL
* No symptomatic pulmonary or visceral Kaposi Sarcoma (KS)

Design:

* Open label, single center pilot Phase II study. Eligible participants receive pacritinib orally 200mg twice daily until progression or up to 6 cycles.
* Participants will be divided by prior therapy for KSHV-MCD (no prior therapy or prior therapy) and by diagnosis of KICS.
* KICS and KSHV-MCD responses will be evaluated by KSHV-MCD Clinical Benefit Response Criteria every 4 weeks.
* Interruptions to pacritinib will be permissible for treatment of worsening KS that develops on study and such interruptions may last up to 12 weeks.
* Radiological assessment using PET-CT and CT will be used to assess response at 1, 3 and 6 months on study.
* Total maximum number of evaluable participants is 54.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must meet KSHV-associated Inflammatory Cytokine Syndrome (KICS) criteria or have histologically or cytologically confirmed Kaposi sarcoma herpesvirus -multicentric Castleman disease (KSHV-MCD) confirmed by the CCR, Laboratory of Pathology (LP), NCI
* Age >= 18 years
* At least one clinical symptom attributed to KSHV-MCD or KICS, as follows:

  * Intermittent or persistent fever for at least 1 week (>38 degrees C)
  * Fatigue (CTCAE - Grade >=2)
  * Gastrointestinal symptoms (e.g., nausea and anorexia - CTCAE Grade >=1)
  * Respiratory symptoms (e.g., cough and airway hyperreactivity - CTCAE Grade >=1)
* At least one laboratory abnormality attributed to KSHV-MCD or KICS, as follows:

  * Anemia (hemoglobin [Hgb] 7.0 - 12.5gm/dL)
  * Thrombocytopenia (50,000 - 150,000/mm3)
  * Hypoalbuminemia (<3.4 g/dL)
  * Elevated C-reactive protein [CRP] (>3mg/L)
* No life or organ-threatening manifestations of KSHV-MCD, KICS or Kaposi Sarcoma (KS)
* Eastern Cooperative Oncology Group [ECOG] performance status <= 3 (Karnofsky >=60%)
* Participants must have laboratory parameters as defined below:

  * Total bilirubin <=3 X upper limit of normal (ULN) or <6X ULN for diagnosis of Gilbert's
  * AST(SGOT)/ALT(SGPT) <=2.5 X ULN
  * PT/PTT/INR <=1.5 X ULN
  * Creatinine within normal institutional limits OR Creatinine clearance >=30mL/min/1.73 m^2 as estimated by either Cockcroft-Gault or 24-hour urine collection for participants with creatinine levels above ULN
* Participants with HIV should be receiving and willing to continue or willing to initiate an effective antiretroviral therapy (ART) regimen that excludes strong/ moderate CYP3A4 inducer or inhibitors.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, participants must be on suppressive therapy.
* Participants with a history hepatitis C virus (HCV) infection must have completed treatment with evidence of sustained virologic response for a period of at least 3 months.
* Participants with KSHV-MCD (Cohort 2) or KICS (Cohort 3) who have received prior therapy, such as rituximab or other monoclonal antibodies, must have a wash out period of at least 3 weeks.
* Participants receiving medications or substances that are substitutes of strong CYP3A4 inhibitors must have a washout period of at least 5 half-lives of the drug prior to enrollment on study.
* Individuals of child-bearing potential (IOCBP) must agree to use a highly effective method of contraception (e.g., intrauterine device [IUD], hormonal [excluding hormonal contraceptives sensitive to CYP3A4 metabolism (i.e. progestin)], surgical sterilization, abstinence) prior to study entry, for the duration of study participation, and for up to 30 days after discontinuation of the study drug.
* Individuals able to father a child with a partner able to become pregnant must agree to use an effective method of contraception (barrier, surgical sterilization, abstinence) for the duration of the study treatment and up to 30 days after the last dose of the study drug.
* Ability of participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Grade >2 symptomatic visceral KS (except for edema or non-ulcerating disease restricted to the oral cavity).
* History of allergic reactions attributed to compounds of similar chemical or biologic

composition to pacritinib.

* Participants receiving any medications or substances that are strong inhibitors or inducers of CYP3A4. Lists including medications and substances known or with the potential to interact with the specified CYP3A4 isoenzymes.
* Participants with evidence of ongoing hemorrhage, active signs/symptoms of bleeding, or history of severe bleeding complications in the one year prior to enrollment.
* Any history of CTCAE grade >= 3 cardiac events within the last 3 months.
* QTc(Fredericia) prolongation >480 ms or other factors that increase the risk for QTc prolongation (i.e., heart failure, or a history of long QT interval syndrome).
* Use of concomitant medications with significant potential for QTc prolongation
* History of thrombosis, troponin-positive (Tpos) or myocardial infarction within the last 6 months
* Participants with moderate (Child-Pugh Score B) or severe hepatic impairment (Child-Pugh Score C)
* Diagnosis of primary effusion lymphoma [PEL] or another lymphoma.
* Participants with a prior or concurrent malignancy whose natural history or treatment that has potential to interfere with the safety or efficacy assessment of the regimen.
* Pregnant individuals as evaluated by a positive serum or urine beta-hCG at screening.
* There is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the nursing person with pacritinib. Breastfeeding should be discontinued if the nursing person is treated with pacritinib.
* Uncontrolled bacterial, mycobacterial, or fungal infection at screening.
* Uncontrolled intercurrent illness that would limit compliance with study requirements, including results of hematology and chemistry testing, infection disease (etc.)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2033-01-01 (Estimated); Study Completion 2034-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit | Prior to each cycle and at EOT and 1 year post treatment
  Percentage of participants with the best overall response of CR or PR to therapy.

SECONDARY OUTCOMES:
Safety of pacritinib | Prior to each cycle, at EOT, and safety visit.
  Adverse events (AEs) will be reported by type and grade of toxicity
Time to treatment failure and duration of benefit | Prior to each cycle and at EOT and 1 year post treatment
  The interval between initiating therapy and the earliest of clinical progression and and the time from to disease progression or death in patients who achieve CR, PR, or SD.
Effect of pacritinib on concurrent diagnosis of Kaposi sarcoma (KS) | Prior to each cycle
  Fraction of participants who have a coexisting diagnosis of KS and who develop a response of any degree (PR; SD)

CONTACTS AND LOCATIONS:
Overall Officials: Ramya M Ramaswami, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested from other researchers after the completion of the primary endpoint.
Access Criteria: Data from this study may be requested by contacting the PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001537-C.html